CLINICAL TRIAL: NCT07403383
Title: Comparative Effects of Strain Counter Strain and Myofascial Release on Pain, Function and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Comparative Effects of Strain Counter Strain and Myofascial Release in Patients With Knee Osteoarthritris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0194
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: pain, quality of life, osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental: Strain Counter Strain (Experimental): Strain Counter Strain involves positioning of hypertonic muscles and dysfunctional joints towards position of comfort. Initial session 2 to 3 times per week. Hot packs 2 to 3 times per week. Tens 2 to 3 times per week. Each session lasts 30 to 60 minutes holding the position for 90 seconds to 2 minutes. Exercises includes.
  Interventions: Other: Strain Counter Strain
- Active Comparator: Myofascial Release (Active Comparator): Myofascial release focuses on the fascia , connective tissue that surrounds muscles, bones and organs which becomes tight and restrict movement. ,Myo fascial release 2 to 3 times per week. 60 seconds per area. Hot packs 2 to 3 times per week. Low frequency TENS. Foam rolling for Calves and Hamstrings. Quadriceps isometric Contraction holds for 10 to 15 seconds with 2 to 4 sets of each exercise. Hamstrings and Adductor isometric contractions.
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Strain Counter Strain — Strain Counter Strain involves passive positioning of hypertonic muscles and dysfunctional joints towards position of comfort. Conventional treatment includes Hot pack, Tens 2 to 3 times per week. Isometric exercises of Quadriceps, Hamstrings, Adductors and Calf muscles
  Arms: experimental: Strain Counter Strain
Other: Myofascial Release — Perform myofascial release technique 2 to 3 times per week. Time 60 seconds per area. Frequency 3 times a week. Hot packs applied 2 to 3 times per week Tens 2 to 3 times per week. Isometric contractions of Quadriceps, Hamstrings , Adductors and Calf muscles hold 10 to 15 seconds then gradually increase 30 seconds with 2 to 4 sets of each exercise
  Arms: Active Comparator: Myofascial Release

SUMMARY:
Osteoarthritis is a degenerative disease, the cartilage present in the joint gets damaged and the bones become hypertrophied. In US, the most commonly occuring arthritis is osteoarthritis. Myofascial release focuses on fascia. Strain counter strain is positional release

ELIGIBILITY:
Inclusion Criteria:

* Both males and females were included in the study.
* Patients aged 40 to 65 with clinical diagnosis of osteoarthritis
* Patient with Grade 2 osteoarthritis
* Patient with Grade 2 osteoarthritis
* Patients who have not undergone any surgical intervention on the Knee in the past 6 months.
* Overweight and obese people with (BMI of 25-29.9), BMI of 30 or above

Exclusion Criteria:

* Patients with history of knee surgery or joint replacement
* Patients with neurological conditions that could affect mobility or perception of pain.
* Patients with infections in the knee area
* Patients with any traumatic injury
* Pregnant Patients

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | at the baseline and at the end of 4 week
  The Numeric Pain Rating Scale is a very common tool to asses pain in clinical settings. It is 0 to 10 pain rating scale in which 0 indicates no pain and 10 indicates worse pain.
Quality of Life (QoL) | at the baseline of 4 weeks
  QoL is 26 item tool has good evidence for reliability, validity and responsiveness to changes in health.

CONTACTS AND LOCATIONS:
Overall Officials: Naila kanwal, TPT, Principal Investigator — Riphah International University
Locations (1):
- PSRD Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No